CLINICAL TRIAL: NCT01456962
Title: Influence of Raltegravir-Containing Antiretroviral Therapy (ART) on Immune Reconstitution and Activation in the Female Genital Tract
Brief Title: Influence of Antiretroviral Regimen on Immune Reconstitution in the Female Genital Tract
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 11-1265; 39423 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2011-10-06; First posted 2011-10-21 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Women's Health; HIV Infection; Genital Diseases, Female
Keywords: Immune reconstitution; CD4+ T cells
MeSH Terms: conditions — HIV Infections; Genital Diseases, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, vaginal fluid samples, cervical biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Raltegravir group: HIV-1-infected women on a regimen of tenofovir (TDF) and emtricitabine (FTC) with raltegravir (RAL)
- Atazanavir group: HIV-1-infected women on a regimen of tenofovir (TDF) and emtricitabine (FTC) with ritonavir (RIT)-boosted atazanavir (ATZ)

SUMMARY:
Increases in cluster of differentiation 4 (CD4)+ T cells in the blood is well documented in human immunodeficiency virus (HIV)-infected individuals after starting antiretroviral therapy (ART), but increases CD4+ T cells in the cervix is variable and not fully understood. Although the amount of HIV in the vagina declines in parallel with those in the plasma when antiretroviral therapy for HIV is started, HIV is still detected frequently in cervical samples from women with undetectable plasma viral loads, suggesting that low level viral replication in the female vaginal tract could lead to both inflammation and incomplete increases in CD4+ T cells. Two classes of HIV medications, nonnucleoside analogue reverse transcriptase inhibitors and protease inhibitors are substantially lower in the female genital tract compared to plasma, whereas concentrations of another class, nucleos(t)ide analogue reverse transcriptase inhibitors are similar or higher to those found in plasma. Thus, many widely used first-line three drug HIV therapies only achieve high concentrations of only two medications in the female genital tract. Importantly, with the recent development of raltegravir (RAL), which achieves concentrations in the female genital tract higher than those in plasma, ART regimens that deliver high concentrations of 3 antiretroviral drugs to the female genital tract are now available. The investigators hypothesize that cervical CD4+ T cell reconstitution is better and inflammatory markers are lower in HIV-infected women on a HIV-therapy including tenofovir (TDF) and emtricitabine (FTC) with RAL versus ritonavir (RIT)-boosted atazanavir (ATZ), and that this is due to therapeutic concentrations of 3 versus 2 antiretroviral drugs in the female genital tract.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive women receiving a RAL-based regimen (n=20) and women receiving an atazanavir-based regimen (n=20).
* Women will be recruited to this study from the Denver metropolitan area.
* The women must have a plasma HIV RNA <48 copies/mL for at least 6 months on the same antiretroviral regimen, and a CD4+ T cell count > 300 cell/mm3.
* Transient increases of <=200 copies HIV-1 RNA copies/ mL will be allowed.

Exclusion Criteria:

* Hysterectomy
* No a menstrual cycle for 12 months
* Active substance abuse
* hematocrit (HCT) <30
* Bleeding diathesis
* Known carcinoma of the cervix
* Using oral glucocorticoids or other immunosuppressive agents
* Current pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1-infected women on a regimen of tenofovir (TDF) and emtricitabine (FTC) with raltegravir (RAL) compared to tenofovir (TDF) and emtricitabine (FTC) and ritonavir (RIT)-boosted atazanavir (ATZ)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Meditz AL, Palmer C, Predhomme J, Searls K, Kerr B, Seifert S, Caraway P, Gardner EM, MaWhinney S, Anderson PL. Relationship Between Genital Drug Concentrations and Cervical Cellular Immune Activation and Reconstitution in HIV-1-Infected Women on a Raltegravir Versus a Boosted Atazanavir Regimen. AIDS Res Hum Retroviruses. 2015 Oct;31(10):1015-22. doi: 10.1089/AID.2014.0301. Epub 2015 Jun 10. PMID 26059647

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir Group: HIV-1-infected women on a regimen of tenofovir (TDF) and emtricitabine (FTC) with raltegravir (RAL) with a CD4+ T-cells/mm3 >300 and HIV RNA copies/mL <48 for a minimum of 6 months.
- Atazanavir Group: HIV-1-infected women on a regimen of tenofovir (TDF) and emtricitabine (FTC) with ritonavir (RIT)-boosted atazanavir (ATZ) with a CD4+ T-cells/mm3 >300 and HIV RNA copies/mL <48 for a minimum of 6 months.
Period: Overall Study
Arm/Group | Raltegravir Group | Atazanavir Group
Started | 16 | 20
Completed | 14 | 19
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir Group | Atazanavir Group | Total
Number analyzed (Participants) | 14 | 19 | 33
Age, Continuous [Mean (Full Range); unit: years] | 44 [31 to 53] | 43 [28 to 65] | 43 [28 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 33
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 19 | 33

OUTCOME MEASURES:

1. Primary Outcome: CD4+ to CD8+ T Cell Ratio in Cervical Biopsies
Description: Evaluation of cervical immune health in HIV-infected women on tenofovir (TDF) and emtricitabine (FTC) and either raltegravir or atazanavir. Cervical CD4+ to CD8+ T cell ratios will be measured at one time point from cervical biopsies. Higher ratios will be a measure of better cervical immune health. In addition, ratios will be compared to the concentration of the drug in the genital tract.
Time Frame: 12 hours after the last medication dose
Measure: Geometric Mean (95% Confidence Interval); unit: Cervical CD4+:CD8+ T cell ratio
Arm/Group | Raltegravir Group | Atazanavir Group
Number analyzed (Participants) | 14 | 19
Cervical CD4+:CD8+ T cell ratio | 0.46 [0.33 to 0.63] | 0.52 [0.36 to 0.75]
Statistical Analysis 1: Comparison: Raltegravir Group vs Atazanavir Group; Test type: Superiority or Other; p = 0.6, t-test, 2 sided
Statistical Analysis 2: Comparison: Raltegravir Group vs Atazanavir Group; Null hypothesis: Higher genital to plasma antiretroviral drug ratios are not associated with higher cervical CD4+:CD8+ T cell ratios; Test type: Superiority or Other; p = 0.4, Regression, Linear; Adjusted for treatment group and time on antiretroviral therapy; % change in CD4+:CD8+ T cells ratio = -9.5, 95% CI 2-sided [-27.3 to 12] — Change based on a 1 log unit increase in genital:plasma drug ratio

ADVERSE EVENTS:
Arm/Group | Raltegravir Group | Atazanavir Group
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/19
Other Adverse Events (participants affected / at risk) | 0/14 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No